CLINICAL TRIAL: NCT01485549
Title: Oligomeric Alpha-synuclein Levels as a Biomarker for Multiple System Atrophy
Brief Title: Oligomeric Alpha-synuclein in Multiple System Atrophy
Acronym: BIOAMS
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2011/11
Record Dates: First submitted 2011-11-29; First posted 2011-12-05 (Estimated); Last update posted 2019-06-27 (Actual); Status verified 2019-02

CONDITIONS: Multiple System Atrophy (MSA)
Keywords: Multiple system atrophy (MSA); alpha-synucleinopathies; biological markers; cerebrospinal fluid; plasma
MeSH Terms: conditions — Multiple System Atrophy; Synucleinopathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * cerebrospinal fluid (CSF)
  * whole blood
  * plasma
  * blood serum
  * urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- MSA Patients: Patients suffering from Multiple system atrophy (MSA)
- Controls: Patients requiring spinal tap without being affected by a neurodegenerative disorder.

SUMMARY:
The main objectives are to determine on one hand whether oligomeric alpha-synuclein levels are increased in MSA patients compared to controls and on other hand whether there is a good agreement between cerebrospinal fluid (CSF) and plasma levels.

DETAILED DESCRIPTION:
Multiple system atrophy (MSA) is a rare neurodegenerative disorder which is characterized by a variable combination of parkinsonism, cerebellar dysfunction, autonomic failure, and additional signs.

No effective treatment is available. Together with PD and Lewy body dementia, MSA belongs to a group of neurodegenerative disorders, the alpha-synucleinopathies, which are characterized by the abnormal accumulation of alpha-synuclein.

The development of biological markers for the diagnosis and prognosis in MSA remains an unmet need. Such biological markers are crucial for future disease-modification and neuroprotection trials. Alpha-synuclein has a high potential for biomarker development since it constitutes the pathological hallmark feature in MSA.

The oligomeric alpha-synuclein seems to be particularly involved in abnormal protein aggregation in alpha-synucleinopathies.

The study will compare alpha-synuclein levels in CSF and plasma between patients suffering from AMS and controls who are patients requiring spinal tap without being affected by a neurodegenerative disorder. The MSA patients and controls will receive CSF and blood sampling at one study visit.

ELIGIBILITY:
* MSA patients

  o Inclusion criteria: Patients suffering from "probable" MSA according to clinical consensus criteria (Gilman et al, 2008), Age >30 Written informed consent Patient covered by the national health system

  o exclusion criteria: UMSARS IV score > 4 points Patient under tutelage Patient unable to give consent Patients receiving anticoagulants, showing abnormal coagulation on blood testing or thrombocytopenia are excluded from this study
* Controls (patients requiring spinal tap without suffering from a neurodegenerative disorder) o Inclusion criteria: Patients not suffering from a neurodegenerative disorder and requiring a spinal tap Age >30 Written informed consent Patient covered by the national health system o exclusion criteria: Similar to MSA patients

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases will be selected from cohort of 90 MSA patients referenced in Bordeaux University Hospital.
  Controls will be selected from patients requiring spinal tap without being affected by a neurodegenerative disorder and paired in age and gender with cases.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2012-11-26 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-11-21 (Actual)

PRIMARY OUTCOMES:
Concentration of oligomeric alpha-synuclein in cerebrospinal fluid (CSF). | Day 0

SECONDARY OUTCOMES:
Total alpha-synuclein concentration in CSF and oligomeric/total alpha-synuclein ratio in CSF | Day 0
Oligomeric and total alpha-synuclein concentration in plasma and oligomeric/total alpha-synuclein ratio in plasma | Day 0
Alpha-synuclein levels in relation to disease duration and age | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Wassilios MEISSNER, MD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Bordeaux University Hospital, Pessac, France